CLINICAL TRIAL: NCT03124667
Title: Cognitive Regulation Training and Exercise (CORTEX)-II With Middle-Aged Adults
Brief Title: Cognitive Regulation Training and Exercise Trial
Acronym: CORTEX-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sean Mullen, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16447; GRANT12053054 (Other Grant/Funding Number: National Institute on Aging); 1R01AG052707-01A1 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-24 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Patient Compliance
Keywords: adherence; cognition; exercise; aging; brain training; cognitive training; executive function
MeSH Terms: conditions — Patient Compliance; Motor Activity | interventions — Games, Experimental; Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gaming Condition (Experimental): The games group will visit the lab on 5 separate occasions, for 2 hours each, to complete training sessions (playing seated and standing computerized games), and then complete 5 similar sessions at home (lasting 2 hours, but may be split into 1-hour sessions at their convenience), at the onset of the exercise program. The training sessions will be scheduled concurrently with exercise classes in the first month. This group will also be asked to accumulate 150 minutes of exercise by attending weekly supervised and unsupervised, group-based aerobic and resistance exercise classes, by visiting the fitness facility alone, and by walking or strength training at home when necessary to supplement fitness facility activities to fully meet public health recommendations, for a period of 12 months.
  Interventions: Behavioral: Games
- Video Condition (Active Comparator): The videos group will visit the lab on 5 separate occasions, for 2 hours each, to view health and educational YouTube videos, and then view 5 similar sessions at home (lasting 2 hours, but may be split into 1-hour sessions at their convenience), at the onset of the exercise program. The training sessions will be scheduled concurrently with exercise classes in the first month. This group will also be asked to accumulate 150 minutes of exercise by attending weekly supervised and unsupervised, group-based aerobic and resistance exercise classes, by visiting the fitness facility alone, and by walking or strength training at home when necessary to supplement fitness facility activities to fully meet public health recommendations, for a period of 12 months.
  Interventions: Behavioral: Videos

INTERVENTIONS:
Behavioral: Games — The game training will emphasize general and exercise-specific dual task processing, self-priming and certainty training.
  Other Names: Gaming Condition
  Arms: Gaming Condition
Behavioral: Videos — The video training will emphasize health and educational information.
  Other Names: Video Condition
  Arms: Video Condition

SUMMARY:
The purpose of this double-blinded, randomized controlled study is to compare CORTEX (Cognitive Regulation Training and Exercise), a multi-faceted, center- and home-delivered- general and exercise-specific-active and traditional computerized cognitive training (CT) program to an attention-control condition involving health and wellness informational videos. More specifically, the cognitive training group will emphasize dual-task abilities, working memory, and visual-spatial processing, as well as self-as-exerciser priming and self-certainty training. It is hypothesized that early intervention cognitive training will enhance use of self-regulatory strategies and self-efficacy and in turn, increase exercise adherence to and engagement in a 12-month aerobic and resistive exercise program at a local fitness facility. More positive improvements in cognitive and psychosocial functioning among participants in the CORTEX condition (relative to the Video Attention-Control condition, i.e., health educational videos), are also expected immediately following the cognitive training, and across time. Expectancies and knowledge of study purpose (blinding integrity) will also be measured and used to statistically adjust for any training differences.

DETAILED DESCRIPTION:
Primary Aim: To test the effectiveness of a 1-month CT (randomized group condition) on exercise self-regulation, a latent factor representing 12-Month exercise adherence & program engagement (i.e., supervised & unsupervised class participation rates, electronically-recorded visitations, Fitbit-derived step counts, & self-reported leisure-time exercise), the investigators will use a structural equation model with robust maximum likelihood estimation. Exercise self-regulation will be regressed on group and known covariates (age, gender, education level, training compliance [percentage of completed sessions], and injury/illness). It is hypothesized that the CORTEX condition will show increased exercise self-regulation (and lower dropout, a categorical outcome variable, tested in a parallel model) compared to the Video Attention-Control condition.

Secondary Aims: A generalized latent variable framework will be used to test the researchers' theorized model and exploratory questions to determine if the CT contributes to greater cognitive change and enhanced perceptions of memory strategy use, self-efficacy, and self-reported physical activity-specific planning and self-regulatory strategy-use; and in turn, greater exercise self-regulation/ lower dropout. To evaluate these questions, first and second-order latent change scores will be derived representing general & exercise-specific cognitive functioning (reaction times and accuracy within training domains), self-efficacy and self-reported self-regulatory strategies, and will be added to the latent exercise self-regulation measurement model (and adjusted with known covariates, i.e., group, age, gender, education, compliance, injury/illness). Positive indirect effects of CT condition on 12-month exercise self-regulation are expected through the change in theoretical constructs-dual task and memory performance, implicit attitudes, memory strategy-use, self-efficacy, exercise planning and physical activity-specific self-regulatory strategy-use. Researchers also predict that the CT program will demonstrate high feasibility/acceptability, as indicated by a thorough process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Low active for the past 3 months
* 35 to 64 years old
* Do NOT regularly play exergames (e.g., XBox Kinect, Playstation Move, Nintendo Wii)
* Do NOT engage in "brain training" regularly (less than once per week)
* Are NOT enrolled in another exercise program or cognitive training study
* Able and willing to comply with the study length, testing, training and exercise program requirements
* Lives within 20 miles of the fitness facility and UIUC research facility
* Has reliable at-home Wi-Fi internet access and an available port for plugging in XBox console
* Vision is at least 20/40 with glasses or contacts with no color blindness
* Do NOT have depression (as defined by a score of 2 or less on the abbreviated Geriatric Depression Scale [GDS-5])
* Do NOT have cognitive impairment (as defined by a score of 21 or higher on the Telephone Interview Cognitive Survey [TICS])

Exclusion Criteria:

* Previously involved in the first CORTEX trial
* Currently involved in regular weekly cognitive training or another physical activity program or study (e.g., yoga, meditation)
* Too active (as defined by regularly exercise 2 or more days per week for 30+ minutes over the past 3 months)
* Incapable of performing moderately intensive aerobic exercise (must be able to complete basic movements, i.e., walking, jogging, jumping, side-stepping, throwing, kicking, punching, grabbing) without exacerbating a pre-existing condition caused by overuse, surgery, or other chronic condition
* Unable or unwilling to comply to lab and home-based training and physical activity prescription
* Unable to commit to full length of program
* Unwilling to be randomized to one of two groups
* Home residence exceeds 20 mile radius from fitness facility or unable to commute to and from fitness facility and UIUC campus
* Do not have reliable at-home Wi-Fi internet access or a required port for plugging in Xbox
* Uncorrectable vision (i.e., less than 20/40 with glasses or contacts with color blindness)
* Depression as defined by GDS >2
* Cognitive impairment as defined by TICS < 21

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 233 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Exercise self-regulation | 12 months
  Exercise self-regulation will be modeled within a latent variable framework. The change factor will be reflected by accumulated supervised and unsupervised class participation rates, total electronically-recorded visitations, averaged monthly Fitbit-derived step counts, and self-reported leisure-time exercise (via Godin Leisure-Time Questionnaire). Measures will be standardized as z-scores. The latent factor model will be adjusted for known covariates (age, gender, education level, training compliance [percentage of completed sessions] and injury/illness) when primary hypothesis of group effects is tested. There is always the possibility that attempts to analyze latent constructs will not converge as planned. In such a case, researchers will attempt to assess change across each behavioral outcome individually with a robust linear regression method, adjusting for multiple comparisons.

SECONDARY OUTCOMES:
Dual task functioning (change) | 1 month
  Four separate heterogeneous dual task transfer assessments will involve auditory and/or visual stimuli. The tasks will progress from a focus on response to singularly-presented stimuli to dual task trials involving equally-prioritized responses (accuracy and quickness) to combinations of colors-letters, pictures-arrows, sounds-voices, and animals-planets. The percentage of incorrect response trials, accuracy, and reaction time will be the outcome measures for each of these tasks. Dual-task percent cost will then be calculated by the following equation: (dual task reaction time - single task reaction time) /single reaction time) x 100. Cost scores will be included as latent factor indicators in a structural equation model testing change from baseline to 1-month follow-up (post-intervention). Measures will be standardized as z-scores.
Memory functioning (change) | 1 month
  Again, from a latent factor perspective, multiple measures will be used to assess the construct of memory functioning, which will reflect overall working memory, spatial and episodic memory. Assessments will be utilized from the iPad-delivered NIH Toolbox, as well computerized assessments developed in E-Prime (e.g., Sternberg). Latent factor memory functioning change from baseline to 1-month follow-up (post-intervention) will be represented by total percent correct for each assessment at each time point. Measures will be standardized as z-scores.
Exercise self-efficacy (change) | 1 month
  Once again, from a latent factor perspective, multiple measures will be used to assess confidence that one can successfully walk longer distances (Self-Efficacy for Walking Scale), continue an exercise regimen (Exercise Self-Efficacy Scale), accumulate physical activity into one's life (Lifestyle Self-Efficacy Scale) and overcome barriers (Barriers Self-Efficacy Scale). An Exercise Self-Efficacy latent factor will be derived from equally-weighted latent factor indicators from each of the scales, and will be used to assess change in exercise-related efficacy beliefs from baseline to 1-month follow-up (post-intervention). Measures will be standardized as z-scores.
Physical activity self-regulatory strategy-use (change) | 1 month
  Participants' perceived use of exercise-specific self-regulatory strategies will be assessed with the multi-dimensional 12-item Physical Activity Self-Regulation Scale. Each of the 12 items will serve as the latent factor indicators for baseline and 1-month follow-up (post-intervention).
Exercise planning (change) | 1 month
  The 10-item Exercise Planning and Scheduling Scale will be used to assess change in exercise-specific planning behaviors from baseline to 1-month follow-up (post-intervention).
Memory strategy-use (change) | 1 month
  Again, from a latent factor framework, multiple self-report scales assessing memory strategy-use (subscale of Metamemory Questionnaire), memory self-efficacy (10-item Memory Self-Efficacy Scale), behavioral self-control (13-item Brief Self-Control Scale), affective and cognitive self-control (10-item Volitional Components Inventory) will be used to derive a latent factor to assess change in perceived Memory Strategy-Use from baseline to 1-month follow-up (post-intervention). Measures will be standardized as z-scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion and after publication of the primary aims and hypotheses, the investigators will provide de-identified data to any interested parties with the provision that they consult with the investigators about the study design, analytical procedures, and to avoid redundancy in future planned analyses or manuscripts. The PI will be given priority and will work closely with other investigators in maximizing ways to leverage the data to address other research questions. Data generated from this project will be made available in multiple formats with codebooks via NCBI's BioProject within 12 months of completing aforementioned priorities. These include demographic information (e.g., age, gender, and education), group assignment codes, and outcome measures. No personally identifying information will be included. Users must also agree to the conditions of use governing access to the public release data.